CLINICAL TRIAL: NCT06946277
Title: Mapping the Temporal Profile of Dexmedetomidine-Induced Analgesia Via EEG Signatures in Brain
Brief Title: Assessing the Time-Course of Dexmedetomidine-Induced Analgesia Via EEG
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China International Neuroscience Institution (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CINI-AD-2025-0218
Record Dates: First submitted 2025-04-11; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Total Hip Arthroplasty (THA); Intrathecal Anesthesia; Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dexmedetomidine Preemptive Analgesia (Experimental)
  Interventions: Drug: Preemptive Analgesia Of Dexmedetomidine

INTERVENTIONS:
Drug: Preemptive Analgesia Of Dexmedetomidine — Preemptive Analgesia Of Dexmedetomidine 1.5 μg · kg-1·h-1 before operation

SUMMARY:
Objective: To investigate the temporal dynamics of dexmedetomidine's analgesic effects in the brain using EEG.

Methods: Eligible patients scheduled for total hip arthroplasty under intrathecal anesthesia received a continuous infusion of DEX at 1.5 μg/(kg·h) for 15 minutes before neuraxial puncture, followed by an additional 15-minute infusion. The study was divided into three phases:

Phase 1: Non-dosing phase (Baseline). Phase 2: DEX preemptive analgesia phase (DEX infusion). Phase 3: DEX cessation phase (Post-infusion).

Outcomes:

Primary safety outcome: EEG spectral analysis at different phases. Secondary outcomes: NRS scores, postoperative nausea and vomiting (PONV), dizziness, agitation, and time to intestinal exhaust within 48 hours. Intraoperative hemodynamics were also monitored.

DETAILED DESCRIPTION:
Objective: To investigate the temporal dynamics of dexmedetomidine's analgesic effects in the brain using EEG.

Methods: Eligible patients scheduled for total hip arthroplasty under intrathecal anesthesia received a continuous infusion of DEX at 1.5 μg/(kg·h) for 15 minutes before neuraxial puncture, followed by an additional 15-minute infusion. The study was divided into three phases:

Phase 1: Non-dosing phase (Baseline). Phase 2: DEX preemptive analgesia phase (DEX infusion). Phase 3: DEX cessation phase (Post-infusion).

Outcomes:

Primary safety outcome: EEG spectral analysis at different phases. Secondary outcomes: NRS scores, postoperative nausea and vomiting (PONV), dizziness, agitation, and time to intestinal exhaust within 48 hours. Intraoperative hemodynamic monitoring was performed.

EEG/ERP monitoring: The 64-site EEG and ERP were recorded at different phases

ELIGIBILITY:
Inclusion Criteria:

Patients with hip osteoarthritis scheduled for total hip arthroplasty under intrathecal anesthesia; Age 18-70 years; American Society of Anesthesiologists (ASA) physical status classification I-III; Body mass index (BMI) 22-30 kg/m².

Exclusion Criteria:

Pre-existing peripheral or central nervous system disorders; Mental disorders; Cognitive impairment; Emergency surgery; or Hearing impairment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-05-26 (Estimated)

PRIMARY OUTCOMES:
Resting EEG | During the whole operation
  Resting-state electroencephalography (rsEEG) was recorded at three phases: before dexmedetomidine infusion (non-dosing phase), during dexmedetomidine infusion (DEX phase), and after dexmedetomidine infusion cessation (Cessation phase).

SECONDARY OUTCOMES:
ERP | During the whole operation
  Event-related potential (ERP) was measured at three phases: before dexmedetomidine infusion (Non-dosing phase), during dexmedetomidine infusion (DEX phase), and after infusion cessation (Cessation phase)

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided